CLINICAL TRIAL: NCT01431755
Title: A Randomised, Subject-blinded Study of Treatment Preference During Cheek Contouring Comparing Restylane® SubQ With and Without the Addition of Lidocaine Hydrochloride 0.3%
Brief Title: A Study of Treatment Preference During Cheek Contouring Comparing Restylane® SubQ With and Without the Addition of Lidocaine Hydrochloride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 31GE1101
Record Dates: First submitted 2011-09-06; First posted 2011-09-12 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2014-04

CONDITIONS: Facial Tissue Augmentation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Restylane SubQ (Other)
  Interventions: Device: Restylane SubQ
- Restylane SubQ Lidocaine (Other)
  Interventions: Device: Restylane SubQ Lidocaine

INTERVENTIONS:
Device: Restylane SubQ — Treatment with up to 2 ml of the product
  Arms: Restylane SubQ
Device: Restylane SubQ Lidocaine — Treatment with up to 2 ml of the product
  Arms: Restylane SubQ Lidocaine

SUMMARY:
The objectives of this study are to evaluate the pain-relieving effect and safety of adding lidocaine hydrochloride to Restylane SubQ and to evaluate the esthetic improvement obtained. The study products will be administered in the cheek.

DETAILED DESCRIPTION:
The Restylane SubQ gel is intended to be used for facial tissue augmentation. The lidocaine content is designed to reduce the subject's pain during treatment. The objectives of this split-face designed study are to evaluate the pain-relieving effect and safety of adding lidocaine hydrochloride to Restylane SubQ and to evaluate the esthetic improvement obtained with the dermal filler using the global esthetic improvement scale (GEIS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Intent to undergo contouring of both cheeks with 1.5 to 2 ml Restylane SubQ per cheek.
* Sufficient symmetry of the face in order to ensure similar volume to be injected, similar injection technique and time for injection.
* Signed informed consent.

Exclusion Criteria:

* Surgery in the midface including aesthetic facial surgical therapy, sinus surgery or dental root surgery within the past 12 months.
* Chronic infection in head and neck region.
* Ongoing infections in mouth.
* Tendency for edema, puffiness or swelling over the zygomatic prominence.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster near or on the area to be treated.
* Previous hypersensitivity to hyaluronic acid or local anesthetics.
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation within 10 days prior to treatment, or a history of bleeding disorders.
* Cancerous or pre-cancerous lesions in the area to be treated.
* Previous tissue augmenting therapy in the area to be treated with non-permanent filler, laser treatment, or chemical peeling during the last 6 months.
* Permanent implant placed in the area to be treated.
* Reduced sensibility in the facial region e.g. due to trauma, facial pareses, previous tissue augmenting therapy, aesthetic facial surgical therapy, laser treatment, or peeling.
* Pregnancy or breast feeding.
* Participation in any other clinical study within 30 days prior to inclusion.
* Other condition preventing the subject to entering the study in the Investigator's opinion e.g. subjects not likely to avoid other facial cosmetic treatments below the level of the upper orbital rim, subjects anticipated to be unreliable or incapable of understanding the VAS assessment, insufficient tissue support or cover of the treatment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedén, M.D., Principal Investigator — Akademikliniken, Storängsvägen 10, 115 42 Stockholm
Locations (3):
- Sweden (3):
  - Plastikkirurggruppen, Stockholm
  - ZMedical, Stockholm
  - Akademikliniken, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: September 10, 2011 Last subject visit: October 19, 2012
Pre-assignment Details: The study has split-face design. Each subject is randomized to treatment with Restylane SubQ in one cheek and Restylane SubQ Lidocaine in the contralateral cheek.
Groups:
- Restylane SubQ/Restylane SubQ Lidocaine: The study has a split-face design. Each subject was injected with Restylane SubQ in one cheek and Restylane SubQ Lidocaine in the contralateral cheek as randomized. Half of the subjects received both study products by injections with a sharp needle and the other half received both study products by injection with a blunt ended microcannula. Following the initial treatment there was a one year follow-up period including an optional re-treatment at 3 months. A maximum volume of 2 ml per cheek and session was recommended.
Period: Overall Study
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Started | 54
Completed | 49
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 3
Region of Enrollment [Number; unit: participants]
  Sweden | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Assessed Treatment With Restylane SubQ Lidocaine as Least Painful.
Description: When injection of both cheeks was completed, the subject was asked which treatment was least painful (right cheek/left cheek/both cheeks alike).
Time Frame: When injection of both cheeks were completed
Population: Intention to treat. 54/54 subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
percentage of participants | 100 [93.4 to 100.0]

2. Secondary Outcome: Subject Pain Assessment by Visual Analogue Scale (VAS) 15 and 120 Minutes After Treatment.
Description: Pain was assessed during the first 2 hours after the initial injection of the study products using a 100 mm VAS. The endpoints of the scale were "no pain" (0 mm) and "worst possible pain" (100 mm). Pain was assessed at the time points 15, 30, 60, 90 and 120 minutes after injection.
Time Frame: 15 and 120 minutes
Population: Intention to treat. 54/54 subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
units on a scale
  Restylane SubQ, VAS at 15 minutes | 28.4 (20.6)
  Restylane SubQ Lidocaine, VAS at 15 minutes | 2.9 (4.1)
  Restylane SubQ, VAS at 120 minutes | 7.3 (11.1)
  Restylane SubQ Lidocaine, VAS at 120 minutes | 1.3 (3.3)

3. Secondary Outcome: Percentage of Improved Subjects at 2 Weeks After Treatment as Assessed by Use of Global Esthetic Improvement Scale (GEIS)
Description: Esthetic improvement was evaluated by using Global Esthetic Improvement Scale. GEIS was evaluated by comparing current photos with pre-treatment photos and using a 5-graded scale (worse/no change/somewhat improved/much improved/very much improved). A clinically significant global esthetic improvement was defined as a score of somewhat improved, much improved or very much improved. GEIS was assessed by the Investigator and the subject. Each cheek/study product was evaluated separately. GEIS was assessed at the time points 2 weeks, 3 months, 2 weeks after re-treatment and 6, 9 and 12 months after first treatment.
Time Frame: 2 weeks
Population: Intention to treat. 54/54 subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
percentage of participants
  Restylane SubQ, subject GEIS, improved | 90.7 [79.7 to 96.9]
  Restylane SubQ, investigator GEIS, improved | 96.3 [87.3 to 99.5]
  Restylane SubQ Lidocain, subject GEIS, improved | 92.6 [82.1 to 97.9]
  Restylane SubQ Lidocaine, invest. GEIS, improved | 100.0 [93.4 to 100.0]

4. Secondary Outcome: Percentage of Subjects With at Least One Step Improvement on Medicis Midface Volume Scale (MMVS) at 2 Weeks
Description: The severity of midface volume loss or midface contour deficiency was assessed by the investigators using a 4-graded scale, Medicis Midface Volume Scale -MMVS (1, fairly full; 2, mild loss of fullness; 3, moderate loss, slight hollowing; and 4, substantial loss, clearly apparent hollowing). Each score were exemplified by photographic images on the scale. A one grade decrease in score from screening was defined as a treatment success/improvement.The efficacy in terms of Medicis Midface Volume Scale (MMVS) was assessed by the Investigator per treatment group. The two cheeks were evaluated separately. MMVS was assessed at the time points 2 weeks, 3 months, 2 weeks after re-treatment and 6, 9 and 12 months after first treatment.
Time Frame: 2 weeks
Population: Intention to treat. 54/54 subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
percentage of participants
  Restylane SubQ, improved MMVS at 2 weeks | 55.6 [41.4 to 69.1]
  Restylane SubQ Lidocaine, improved MMVS at 2 weeks | 59.3 [45.0 to 72.4]

5. Secondary Outcome: Number of Subjects Reporting at Least 1 Diary Complaint Related to the Cheek Treated With Restylane SubQ and Restylane SubQ Lidocaine Respectively After Initial Treatment.
Description: A subject diary was completed for 14 days following the initial treatment and the optional re-treatment at the 3-month visit. Each subject was asked to record the presence of bruising, redness, swelling, pain, tenderness and itching.
Time Frame: 14 days
Population: Safety Population. 54/54 subjects.
Measure: Number; unit: participants
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
participants
  Restylane SubQ | 54
  Restylane SubQ Lidocaine | 52

6. Secondary Outcome: Number of Subjects Reporting Adverse Event
Description: Adverse Events (AEs) were collected by open questioning, information obtained from signs and symptoms detected during examination, observed by the study personnel or spontaneous reports from the subjects.
  All subjects were injected with Restylane SubQ in one cheek and Restylane SubQ Lidocaine in the contralateral cheek.
Time Frame: Up to 12 months
Population: Safety population, 54 subjects.
Measure: Number; unit: participants
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine
Number analyzed (Participants) | 54
participants | 41

ADVERSE EVENTS:
Time Frame: From treatment up to 12 months
Description: Adverse Events (AEs) were collected by open questioning, information obtained from signs and symptoms detected during examination, observed by the study personnel or spontaneous reports from the subjects.
Groups:
- Restylane SubQ/Restylane SubQ Lidocaine: Systemic; Restylane SubQ: Localized; Restylane SubQ Lidocaine: Localized: The study has a split-face design. Each subject was injected with Restylane SubQ in one cheek and Restylane SubQ Lidocaine in the contralateral cheek as randomized. Half of the subjects received both study products by injections with a sharp needle and the other half received both study products by injection with a blunt ended microcannula. Following the initial treatment there was a one year follow-up period including an optional re-treatment at 3 months. A maximum volume of 2 ml per cheek and session was recommended.Hence, all subjects received injections with both products at the same time.
Arm/Group | Restylane SubQ/Restylane SubQ Lidocaine: Systemic | Restylane SubQ: Localized | Restylane SubQ Lidocaine: Localized
Serious Adverse Events (participants affected / at risk) | 4/54 | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 9/54 | 25/54 | 20/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane SubQ/Restylane SubQ Lidocaine: Systemic (N=54) | Restylane SubQ: Localized (N=54) | Restylane SubQ Lidocaine: Localized (N=54)
Mesenteric Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic Ulcer Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane SubQ/Restylane SubQ Lidocaine: Systemic (N=54) | Restylane SubQ: Localized (N=54) | Restylane SubQ Lidocaine: Localized (N=54)
Implant site inflammation (General disorders) | 0 (0) | 11 (30) | 10 (21) — All subjects recovered from these reaction before study end.
Implant site swelling (General disorders) | 0 (0) | 6 (7) | 5 (5)
Injection site pain (General disorders) | 0 (0) | 9 (9) | 4 (4)
Implant site nodule (General disorders) | 0 (0) | 7 (7) | 4 (4)
Implant Site Pruritus (General disorders) | 0 (0) | 3 (4) | 4 (7)
Implant site erythema (General disorders) | 0 (0) | 3 (3) | 3 (3)
Implant site haematoma (General disorders) | 0 (0) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or presentation by PI shall be submitted to Q-Med for review no less than 60 days before submission for publication or presentation. Q-Med will provide any comments to Principal Investigator within thirty (30) days following receipt of the proposed publication/presentation. PI agrees to consider, discuss and give reasonable considerations to comments by Q-Med. Q-Med may also request that the Company name or Q-Med employee name appear or not appear in such publication.